CLINICAL TRIAL: NCT06321081
Title: ICE Study: a Clinical Study of the Combination of Irinotecan Plus Cetuximab and Envafolimab as a Rechallenge Regimen in mCRC
Brief Title: ICE Study: Combination of Irinotecan Plus Cetuximab and Envafolimab as a Rechallenge Regimen in mCRC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Hospital (Other Government)
Collaborators: Bethune Charitable Foundation (Unknown)
Responsible Party: Principal Investigator, Yingying Huang, investigator, Beijing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023BJYYEC-428-02
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: RAS Mutation; Metastatic Colorectal Cancer; MSS
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Cetuximab; envafolimab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICE treatment group (Experimental): any RAS wild type mCRC patients who had got benefits from cetuximab or irinotecan will be treated with ICE regimen (Irinotecan 150mg/m2,Q2W, cetuximab 500mg/m2, Q2W, envafolimab 200mg, Q2w)
  Interventions: Drug: irinotecan, cetuximab, envafolimab

INTERVENTIONS:
Drug: irinotecan, cetuximab, envafolimab — rechallenge treatment
  Other Names: CPT-11, PD-L1 inhibitor

SUMMARY:
This is a non-profit phase II, open, clinical study of the combination of irinotecan plus cetuximab and envafolimab as a rechallenge regimen, in pre-treated RAS/BRAF wild type metastatic colorectal cancer patients (according to liquid biopsy at baseline). Patients have been treated in front lines with irinotecan and cetuximab and had a clinical benefit (complete or partial response) from both of them, no matter whether they had treated by any PD-1 inhibitor before.

DETAILED DESCRIPTION:
This is a non-profit phase II, open-label, clinical study of the combination irinotecan plus cetuximab and envafolimab as a rechallenge regimen, in pre-treated RAS/BRAF wild type metastatic colorectal cancer patients (according to liquid biopsy at baseline). Patients have been treated in front lines with irinotecan and cetuximab and had a clinical benefit (complete or partial response) from both of them, no matter whether they had treated by any PD-1 inhibitor before.

30 patients will be treated with irinotecan plus cetuximab and envafolimab. For each patient, before treatment, a blood sample will be obtained and analyzed for circulating free tumorDNA, to identify RAS/BRAF wild type patient to be enrolled.

The same procedure will be performed at progression of the disease. Treatment will continue until:

disease progression. significant clinical deterioration any criterion for withdrawal from the trial or trial drug is fulfilled treatment may continue past the initial determination of disease progression according to RECIST 1.1. if the subject's performance status has remained stable, and if in the opinion of the Investigator, the subject will benefit from continued treatment and if other criteria are fulfilled as outlined in the protocol, that is, no new symptoms or worsening of existing symptoms and no decrease in performance score.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent before any trial-related procedure is undertaken that is not part of the standard patient management.

Male or female subjects aged ≥ 18 years. Histologically proven diagnosis of colorectal adenocarcinoma. Diagnosis of metastatic disease. RAS (NRAS and KRAS exon 2,3 and 4) and BRAF wild-type in liquid biopsy at screening (according to NGS) Efficacy of any front-line therapies containing cetuximab or irinotecan with a major response achieved (i.e. complete or partial response according to RECIST criteria v1.1)..

More than 2 months since the last dose of cetuximab administered in first line treatment before randomization.

Measurable disease according to RECIST criteria v1.1. ECOG PS of 0 to 1 at trial entry. Estimated life expectancy of more than 12 weeks. Adequate hematological function defined by white blood cell (WBC) count ≥ 2.5 × 109/L with absolute neutrophil count (ANC) ≥ 1.5 × 109/L, lymphocyte count ≥ 0.5 × 109/L, platelet count ≥ 100 × 109/L, and hemoglobin ≥ 9 g/dL (may have been transfused).

Adequate hepatic function defined by a total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range and AST and alanine aminotransferase (ALT) levels ≤ 2.5 × ULN for all subjects or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver).

Adequate renal function defined by an estimated creatinine clearance > 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method).

Effective contraception for both male and female subjects throughout the study and for at least 2 months after last study treatment administration if the risk of conception exists (Note: The effects of the trial drug on the developing human fetus are unknown; thus, women of childbearing potential and men must agree to use effective contraception, defined as 2 barrier methods, or 1 barrier method with a spermicide, an intrauterine device, or use of oral female contraceptive. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this trial, the treating physician should be informed immediately).

Exclusion Criteria:

* Any contraindication to cetuximab and/or envafolimab. Past or current history of malignancies other than colorectal carcinoma, except for curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix.

Pregnancy. Breastfeeding. Participation in a clinical study or experimental drug treatment within 30 days before enrollment.

Subjects receiving immunosuppressive agents (such as steroids) for any reason, should be tapered off these drugs before initiation of the trial treatment, with the exception of:

Subjects with adrenal insufficiency, who may continue corticosteroids at physiologic replacement dose, equivalent to ≤ 10 mg prednisone daily Intranasal, inhaled, topical steroids, Local steroid injection (e.g., intra-articular injection) Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) No ongoing neurological symptoms related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable) Prior organ transplantation, including allogeneic stemcell transplantation

Significant acute or chronic infections including, among others:

Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome

Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent:

Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.

Subjects requiring hormone replacement with corticosteroids are eligible if steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or equivalent prednisone per day.

Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) are acceptable.

Active infection requiring systemic therapy. Previous or ongoing administration of systemic steroids for the management of an acute allergic phenomenon is acceptable as long as it is anticipated that the administration of steroids will be completed in 14 days, or that the daily dose after 14 days will be ≤ 10 mg per day of equivalent prednisone.

Known severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v 5 Grade ≥ 3), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma).

History of hypersensitivity to Polysorbate 80 that led to unacceptable toxicity requiring treatment cessation.

Persisting toxicity related to prior therapy of Grade > 1 NCI- CTCAE v 5.0. Known alcohol or drug abuse. Clinically significant (that is active) cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class ≥ II), or serious uncontrolled cardiac arrhythmia requiring medication.

History of keratitis, ulcerative keratitis or severe dry eye. Since contact lent use is also a risk factor for keratitis and ulceration, it is not recommended.

Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Legal incapacity or limited legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-08-14 (Estimated)

PRIMARY OUTCOMES:
progression free survival | from screening up to 36 months (from the start of therapy until disease progression or death due to any cause
  the interval from enrollment to disease progression

SECONDARY OUTCOMES:
Overal survival | from screening up to 36 months (from the start of therapy until death due to any cause
  the interval from enrollment to death for every cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided